CLINICAL TRIAL: NCT03353025
Title: Prospective Randomized Clinical Study on Transsphenoidal or Dopamine Drugs Therapy Treat Non-invasive Prolactinoma
Brief Title: Study on Therapy of Non-invasive Prolactinoma
Acronym: TNAPA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Hai-Jun Wang, director, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016008
Record Dates: First submitted 2017-02-20; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Prolactinoma
Keywords: non-invasive prolactinoma
MeSH Terms: conditions — Prolactinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transsphenoidal surgery treatment (Experimental): Transsphenoidal surgery treat non-invasive prolactinoma by experienced neurosurgeon
  Interventions: Procedure: transsphenoidal surgery treatment
- dopamine agonist treatment (Experimental): Minimum effective dose of dopamine agonist, bromocriptine, treat non-invasive prolactinoma
  Interventions: Drug: dopamine agonist treatment

INTERVENTIONS:
Procedure: transsphenoidal surgery treatment — transsphenoidal surgery treatment
  Other Names: TSS
  Arms: transsphenoidal surgery treatment
Drug: dopamine agonist treatment — Minimum effective dose of dopamine agonist，bromocriptine，treat prolactinona
  Other Names: DA
  Arms: dopamine agonist treatment

SUMMARY:
the study aim to investigate the endocrine remission rate of non-invasive prolactinoma between transsphenoidal surgery treatment and Dopamine agonist treatment.

DETAILED DESCRIPTION:
Non-invasive prolactinomas were treated by transsphenoidal surgery or Dopamine agonist until now. However，this two type therapies were controversial. The study aim to investigate the endocrine remission rate of non-invasive prolactinoma between transsphenoidal surgery treatment and Dopamine agonist treatment.

ELIGIBILITY:
Inclusion Criteria:

non-invasive prolactionma

Exclusion Criteria:

invasive prolactioma

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 394 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Endocrine remission rate | five-year
  After intervention, blood prolactin normalization rate

CONTACTS AND LOCATIONS:
Overall Officials: Haijun Wang, Dr., Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Sun Yat-sen 5010 program, Guangzhou, China